CLINICAL TRIAL: NCT06977438
Title: Promoting Healthy Children and Youth
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2025-33936
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- High Dose HBLT (Experimental): Individuals in this group will be randomized in an open fashion to receive 26 hours of HBLT during the course of the study. Participants will have HBLT every two weeks during the study which will entail 45 minute virtual group classes with a 15 minute individual goal setting session.
  Interventions: Drug: Semaglutide
- Medium Dose HBLT (Experimental): Individuals in this group will be randomized in an open fashion to receive 13 hours of HBLT during the course of the study. Participants will have HBLT every four weeks during the study which will entail 45 minute virtual group classes with a 15 minute individual goal setting session.
  Interventions: Drug: Semaglutide
- Low Dose HBLT (Experimental): Individuals in this group will be randomized in an open fashion to receive 4 hours of HBLT during the course of the study. Participants will have HBLT at four timepoints during the study (Weeks 2, 18, 34 and 50) which will entail 45 minute virtual group classes with a 15 minute individual goal setting session.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — All participants in this study will receive treatment with Semaglutide

SUMMARY:
The rapid emergence of new and highly effective obesity medications has turned the field of pediatric weight management on its head. Adolescents living with obesity, their caregivers, healthcare providers, healthcare systems, policymakers, and payors are now wondering what role health behavior and lifestyle treatment (HBLT) has in terms of body mass index (BMI) reduction, improvements in quality of life and cardiometabolic health, and mitigating nutritional concerns when medications are used. Is intensive (26+ hours) of HBLT needed or could low intensity HBLT be an equally effective alternative; and if so, for whom? Our proposed project will answer these important questions that arise daily in the clinical setting and will generate critical new insights to guide decision-making for teens with obesity and the stakeholders who care deeply about them.

DETAILED DESCRIPTION:
The premise underpinning our proposed project stems from the conceptual framework that obesity medications beneficially alter the underlying pathophysiology that largely drives eating behaviors (appetite, satiety, cravings, and "food noise"), thereby lessening the need for high doses of HBLT. In this way, medications can unburden adolescents living with obesity, their caregivers, healthcare providers, health systems, and payors from the need to engage in and provide intensive HBLT. This framework has directly informed our research strategy and methodological approach, including the design of our trial and the variables we have chosen to assess. Indeed, we plan to compare three different doses of HBLT in terms of their ability to improve health-related outcomes while having a keen eye on nutritional safety and eating disorders. The design and patient-centered outcomes for our trial have been carefully and thoughtfully crafted to provide evidence-based clarity on critical decisional dilemmas regarding how much HBLT is needed to get the most out of obesity pharmacotherapy and how social determinants of health (SDOH) factors can help guide treatment strategies to maximize effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to < 18 years at screening
* BMI >/= 95th percentile based on age and sex

Exclusion Criteria:

* Diabetes (type 1 or 2) due to safety concerns about properly surveiling glycemic control virtually
* Current or recent (< 6 months prior to screening) use of obesity medications
* Previous metabolic/bariatric surgery
* Current or recent (< 6 months prior to screening) use of medication(s) to treat insulin resistance
* Hypertension
* Hypercholesterolemia
* History of treatment with growth hormone
* Eating disorder diagnosis
* Major psychiatric disorder
* Unstable clinically-diagnosed depression
* History of suicide attempt
* History of suicidal ideation or self-harm within 30 days of screening
* Current pregnancy or plans to become pregnant
* Tobacco use
* Uncontrolled hypertension
* Diagnosis of monogenic obesity
* History of cholelithiasis without cholecystectomy
* Untreated thyroid disorder
* History of pancreatitis
* Personal/family history of medullary thyroid carcinoma and/or multiple endocrine neoplasia type 2

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1020 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2031-01-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) Reduction | 24 months
  Change in body mass index

IPD SHARING:
Plan to Share IPD: Undecided